CLINICAL TRIAL: NCT07062328
Title: Efficacy and Safety of Recaticimab (PCSK9 Inhibitor) and Adebrelimab Combined With Chemotherapy as First-line Treatment for Unresectable/ Advanced Biliary Tract Carcinoma: A Single-arm, Phase II Study
Brief Title: A Trial of Recaticimab and Adebrelimab in Combination With Chemotherapy in Patients With Unresectable BTC
Acronym: HP-BTC-002
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dong sheng Zhang, Chief physician，professor, Sun Yet-Sen University Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2025-251-02
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Carcinoma
Keywords: GP chemotherapy; Antineoplastic Agents; PCSK9 Inhibitor; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Recaticimab and Adebrelimab in Combination With chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recaticimab and Adebrelimab in Combination With chemotherapy (Experimental): Adebrelimab (SHR-1316) is a novel humanised IgG4 monoclonal antibody against PD-L1.
  Recaticimab is a new humanized IgG1 monoclonal antibody developed to selectively target PCSK9 with the potential for durable action.
  Interventions: Drug: Recaticimab and Adebrelimab; Drug: GP chemotherapy

INTERVENTIONS:
Drug: Recaticimab and Adebrelimab — Patients would receive Recaticimab (150 mg, sc., q4w) and Adebrelimab (1200 mg, iv., q3w) plus GP chemotherapy in 21day cycles.
  Recaticimab and Adebrelimab would be maintained until the disease progressed or intolerable toxicity and adverse reactions or the medication was used for two years.
Drug: GP chemotherapy — Gemcitabine/Cisplatin (gemcitabine 1000mg/m2 + cisplatin 25mg/m2) will be administered on D1/D8 in every three weeks cycle, up to 6 cycles.

SUMMARY:
The study aims to evaluate the efficacy and safety of Recaticimab and Adebrelimab in Combination With chemotherapy in patients with metastatic biliary tract carcinoma (BTC).

DETAILED DESCRIPTION:
The investigators are conducting a clinical research study to evaluate the effectiveness and safety of a novel combination therapy for patients with advanced, unresectable biliary tract carcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1. Provided informed consent and sign the informed consent form;
* 2. Male or female, Aged 18-75 years (counted on the date of signing informed consent);
* 3. Histologically confirmed unresectable advanced or metastatic biliary tract adenocarcinoma, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma.;
* 4. The patient is not a candidate for surgery, or the disease has progressed after prior surgery and/or local treatment.
* 5. No previous systematic treatment for advanced BTC. Exceptions include patients who relapsed more than 6 months after adjuvant chemotherapy following radical resection. Local regional therapy (including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic arterial infusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) must have been completed at least 4 weeks prior to baseline radiological scanning, and any toxicity (except alopecia) induced by local regional therapy must have resolved to ≤ Grade 1 in accordance with National Cancer Institute - Common Terminology Criteria for Adverse Event version 5.0 (NCI-CTCAE v5.0);
* 6. No prior treatment with immune-mediated therapy, including but not limited to other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, with the exception of therapeutic anticancer vaccines and adjuvant immunotherapy administered after curative resection
* 7. Have at least one measurable lesion (in accordance with RECIST v1.1, major diameter ≥ 10 mm of the measurable lesion in spiral CT scan or short diameter of swollen lymph node ≥ 15 mm; the lesion with previous local therapy can be used as target lesion after the progression is confirmed in accordance with RECIST v1.1)
* 8. Child-Pugh class: Grade A
* 9. ECOG-PS score: 0-1;
* 10. With a life expectancy of ≥ 12 weeks;
* 11. Adequate major organ function without severe hematologic, cardiac, pulmonary, hepatic, renal, or bone marrow dysfunction, and no immunodeficiency disease;
* 12. For active hepatitis B, it is required that effective antiviral treatment be received (according to local standard therapy, such as entecavir or tenofovir), with HBV DNA ≤ 2000 IU/mL or a reduction of HBV DNA by 10 times after antiviral treatment, and the patient must agree to continue effective anti-HBV treatment throughout the study period;
* 13. Women of childbearing potential must agree to abstain from heterosexual intercourse or use reliable contraception from the time of signing informed consent until at least 120 days after the last study drug administration. A negative serum pregnancy test (HCG) must be confirmed within 7 days before starting study treatment. Lactating women are excluded;
* 14. Men with female partners of childbearing potential must agree to abstain from heterosexual intercourse or use reliable contraception from the time of signing informed consent until at least 120 days after the last study drug administration. Men must also agree not to donate sperm during this period. For men whose partners are pregnant, condom use is required without additional contraception;

Exclusion Criteria:

* 1. Other active malignant tumor exceptBTCwithin 5 years or simultaneously. Cured localized tumor, for example, basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate, carcinoma in situs of cervix, breast cancer in situ may be enrolled;
* 2. A previous diagnosis of nephrotic syndrome, severe liver disease, Cushing's syndrome, or other diseases that significantly affect lipid levels; a history of low cholesterol, low lipidemia, or related family history, or a family history of allergy to PCSK inhibitors
* 3. Planning to or previously received organ or allogenic bone marrow transplantation;
* 4. Treatment of other investigational product(s) within 28 days prior to the start of study treatment;
* 5. Moderate or severe ascites with clinical symptoms that require therapeutic puncture and drainage, or Child-Pugh score >2 (excluding those with only a small amount of ascites on imaging without accompanying clinical symptoms); uncontrolled or moderate to large pleural effusion, pericardial effusion;
* 6. History of gastrointestinal bleeding within 6 months prior to the start of study treatment or clear tendency of gastrointestinal bleeding;For example, those with a risk of bleeding or severe esophageal and gastric varices, active local gastrointestinal ulcer lesions, persistent positive fecal occult blood test cannot be enrolled (if the fecal occult blood test is positive at baseline, it can be rechecked. If it remains positive after re-examination, an endoscopy (EGD) should be performed. Those who are found to have esophageal and gastric varices with a high risk of bleeding by EGD cannot be enrolled);
* 7. Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment
* 8. Known genetic or acquired hemorrhage (e.g., coagulation dysfunction) or thrombotic tendency, for example, subject with hemophilia; current or recent (within 10 days prior to the start of study treatment) use of full-dose of oral or intravenous anticoagulant or thrombolytic drug for the purpose of treatment (preventive use of low-dose aspirin or low molecular weight heparin is allowed);
* 9. Current or recent (within 10 days prior to the start of study treatment) use of aspirin (> 325 mg/day, maximum dose for antiplatelet) or dipyridamole, ticlopidine, clopidogrel and cilostazol;
* 10. Thrombosis or thromboembolic event within 6 months prior to the start of study treatment, for example, cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism;
* 11. Cardiac clinical symptom or disease that is not well controlled;
* 12. Hypertension that cannot be well controlled through antihypertensive drugs, allowing to reach the above parameters by the use of antihypertensive therapy; previous hypertensive crisis or hypertensive encephalopathy;
* 13. Major vascular disease within 6 months prior to the start of study treatment (for example, aortic aneurysm requiring surgical repair or peripheral arterial thrombosis in recent days); Serious, unhealed or splitting wound and active ulcer or untreated bone fracture; Major surgical therapy within 4 weeks prior to the start of study treatment (except diagnosis), or planned major surgery during the study;
* 14. Evidence on intraperitoneal pneumatosis that can not be explained by puncture or recent surgery;
* 15. Previous or current presence of metastasis to central nervous system; Metastatic disease involving main airway or blood vessels (e.g. Vena cava tumor invasion or complete occlusion of the major portal vein due to HCC, the major portal vein is defined as the part of portal vein between the union of the splenic and superior mesenteric veins and the first bifurcation into the left and right vein) or high-volume mediastinal tumor mass located in the center (distance from carina <30 mm);
* 16. History of hepatic encephalopathy; Current interstitial pneumonia or interstitial lung disease, or history of interstitial pneumonia or interstitial lung disease which required hormonal therapy, or other pulmonary fibrosis that may interfere with the judgement and treatment of immune-related pulmonary toxicity; organizing pneumonia (e.g., obliterative bronchiolitis), pneumoconiosis, drug related pneumonitis, idiopathic pneumonia, subjects with evidence on active pneumonia or serious pulmonary function impairment on thoracic computed tomography (CT) in screening period (previous radiation pneumonitis in the radiation area will be allowed); active tuberculosis;
* 17. Active autoimmune disease or history of autoimmune disease and may relapse (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [with the exception that it can be controlled by hormone replacement therapy]). Subjects with skin disease that do not require systemic treatment are eligible, for example, leukoderma, psoriasis, alopecia; subjects with controlled type 1 diabetes by insulin are eligible; subjects with asthma that has been completely resolved in childhood and don't need any treatment are eligible, but subjects with asthma that require a bronchodilator as medical intervention are not eligible;
* 18. Use of immunosuppressive medication within 14 days prior to the start of study treatment, or systemic corticosteroid therapy to achieve the objective of immunosuppression (Prednisone at the dose of >10mg/day or equivalent);
* 19. Known history of hypersensitivity to the active substance or to any other components of each investigational medicinal product;
* 20. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia or complications of severe pneumonia; oral or intravenous therapeutic antibiotics within 2 weeks prior to the start of study treatment (subjects who are treated with antibiotics for prevention, e.g., preventive urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible for participation in the study);
* 21. Congenital or acquired immunodeficiency (e.g., HIV infection);
* 22. Hepatitis B and hepatitis C co-infection;
* 23. Attenuated live vaccine therapy administered within 28 days prior to the start of study treatment, or are expected to receive such vaccines during Adebrelimab treatment or within 60 days after the last dose of Adebrelimab;
* 24. Other factors that may affect the study results or lead to early study termination as judged by investigators, such as alcoholism, drug abuse, other serious diseases (including mental disorders) requiring concomitant therapy, with serious laboratory examination abnormality, with family or social factors, that may affect subject's safety.
* 25.Other conditions in which the investigator deems the subject unsuitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | up to 24 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Progression-Free Survival (PFS) | up to 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Adverse Events (AE) | up to 24 months
  Overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

IPD SHARING:
Plan to Share IPD: No